CLINICAL TRIAL: NCT06641609
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antitumor Activity of CFT8919 Capsules in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC).
Brief Title: A Phase I Study of CFT8919 in Patients With Advanced NSCLC
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTP-662212
Record Dates: First submitted 2024-09-20; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Non-Small Cell Lung Cancer With EGFR Mutation
Keywords: Non-small cell lung cancer; EGFR mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose-Escalation (Phase Ia) (Experimental): Intervention Name: CFT8919 capsule Intervention Type: Drug Intervention Description: Participants will receive CFT8919 at different dose levels in a "3+3" dose-escalation design, starting from 150 mg BID, increasing to 300 mg, 600 mg, and up to 900 mg BID.
  Interventions: Drug: Dose-Escalation (Phase Ia) CFT8919 capsule
- Dose-Expansion (Phase Ib) (Experimental): After the MTD is determined in Phase Ia, participants will receive CFT8919 at the recommended Phase II dose (RP2D). The primary objective is to further evaluate the safety and preliminary antitumor activity of the drug at the RP2D
  Interventions: Drug: Dose-Expansion (Phase Ib) CFT8919 capsule
- Cohort-Expansion (Phase Ic) (Experimental): Participants will be enrolled based on their EGFR mutation status into separate cohorts. Each cohort will receive CFT8919 at the RP2D to evaluate its efficacy, safety, and pharmacokinetic profile in specific EGFR mutation populations, including those with L858R and other EGFR-resistant mutations after EGFR-TKI treatment.
  Interventions: Drug: Cohort-Expansion (Phase Ic) CFT8919 capsule

INTERVENTIONS:
Drug: Dose-Escalation (Phase Ia) CFT8919 capsule — Phase 1a，enrolled, eligible patients receive CFT8919 150-900mg twice daily.
  Other Names: CFT8919
  Arms: Dose-Escalation (Phase Ia)
Drug: Dose-Expansion (Phase Ib) CFT8919 capsule — Phase 1b，enrolled, eligible patients receive CFT8919 RP2D twice daily.
  Other Names: CFT8919
  Arms: Dose-Expansion (Phase Ib)
Drug: Cohort-Expansion (Phase Ic) CFT8919 capsule — Phase 1c，enrolled, eligible patients receive CFT8919 RP2D twice daily.
  Other Names: CFT8919
  Arms: Cohort-Expansion (Phase Ic)

SUMMARY:
The goal of this clinical trial is to evaluate the safety, tolerability, pharmacokinetics, and antitumor activity of CFT8919 capsules in patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) carrying EGFR mutations. The main questions it aims to answer are:

* What is the maximum tolerated dose (MTD) of CFT8919?
* Does CFT8919 demonstrate antitumor activity in these patients?

Participants will:

* Take CFT8919 capsules at different doses.
* Undergo regular assessments for safety, pharmacokinetics, and tumor response. Researchers will compare different dose levels to determine the best balance between safety and efficacy.

DETAILED DESCRIPTION:
This is a Phase I clinical study designed to evaluate the safety, tolerability, pharmacokinetics, and antitumor activity of CFT8919 capsules in patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) who carry EGFR mutations. The study includes three parts: dose-escalation, dose-expansion, and cohort-expansion. The primary objectives are to determine the maximum tolerated dose (MTD) in the dose-escalation phase and to assess the antitumor efficacy in the cohort-expansion phase. Secondary objectives include assessing pharmacokinetic parameters, objective response rate (ORR), disease control rate (DCR), progression-free survival (PFS), and overall survival (OS). Exploratory objectives will evaluate biomarkers and the relationship between drug exposure and treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Dose-Escalation and Dose-Expansion Phases: Patients with histologically or cytologically confirmed locally advanced or metastatic non-small cell lung cancer (NSCLC) harboring the EGFR-L858R mutation, who have failed standard treatment (disease progression or intolerance), lack standard treatment options, or are deemed unsuitable for standard treatment by the investigator, or have refused standard treatment.
2. Cohort-Expansion Phase: In addition to the above criteria, the following must also be met:

   * Cohort A: Patients with locally advanced or metastatic NSCLC harboring the EGFR-L858R mutation who have experienced disease progression after third-generation EGFR-TKI treatment and carry secondary EGFR mutations (such as C797S, L718Q, G724S, S768I, etc.).
   * Cohort B: Patients with locally advanced or metastatic NSCLC harboring the EGFR-L858R mutation who have failed standard treatment or are unsuitable for or have refused standard treatment (patients with secondary EGFR mutations are prioritized for Cohort A).
3. • Dose-Escalation Phase requires evaluable lesions, while Dose-Expansion and Cohort-Expansion Phases require measurable lesions as defined by RECIST V1.1.
4. • Age ≥18 years, no gender restrictions.
5. • Expected survival ≥12 weeks.
6. • Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
7. • Adequate organ function, meeting the following criteria:

   * Hematologic: Absolute neutrophil count (ANC) ≥1.5 × 10⁹/L (1500/mm³), platelets ≥100 × 10⁹/L, hemoglobin ≥9 g/dL (90 g/L) without transfusion or hematopoietic growth factors within 14 days prior to screening.
   * Coagulation: International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤1.5 × the upper limit of normal (ULN).
   * Liver: Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 × ULN, or ≤5.0 × ULN in the presence of liver metastases; total bilirubin (TBIL) ≤1.5 × ULN, or ≤3.0 × ULN in the presence of liver metastases or known Gilbert's syndrome (unconjugated hyperbilirubinemia).
   * Kidney: Serum creatinine (Scr) ≤1.5 × ULN, or for patients with Scr >1.5 × ULN, creatinine clearance (Ccr) ≥50 mL/min (calculated using the Cockcroft-Gault formula); urine protein ≤1+, or if ≥2+, 24-hour urine protein quantification showing <1 g.
8. • Toxicity from prior anti-tumor treatments must have resolved to CTCAE grade ≤1 (except for toxicities that, in the investigator's judgment, are long-lasting and non-recoverable but pose no safety risk and are ≤2 in grade).
9. • Patients must have been previously diagnosed with the EGFR-L858R mutation via local testing. In the Dose-Escalation and Dose-Expansion Phases, patients who progressed on prior EGFR-TKI treatment must provide the genetic mutation results from their most recent EGFR-TKI treatment. For Cohort A patients, progression on third-generation EGFR-TKI treatment must have confirmed the presence of secondary EGFR mutations (e.g., C797S, L718Q, G724S, S768I) via tissue or blood tests.
10. • Patients must be willing to provide blood samples and optionally provide tissue samples for exploratory biomarker research.
11. • Non-breastfeeding women of childbearing potential must have a negative serum or urine pregnancy test within 7 days before starting study treatment, and all enrolled patients must agree to use medically accepted contraception for 1 month prior to treatment, during the entire treatment period, and for 3 months after completing treatment.
12. • Signed informed consent form.

Exclusion Criteria:

1. Prior or ongoing treatment with EGFR-L858R-targeted PROTAC therapies.
2. Less than 5 half-lives or 4 weeks (whichever is shorter) since the last anti-tumor treatment before the first dose of study drug; less than 6 weeks since the last treatment with nitrosoureas or mitomycin C; less than 1 week since the last anti-tumor herbal treatment.
3. Patients who underwent major surgery (as defined by the investigator) or experienced significant trauma within 4 weeks before the first dose of study drug; patients who received radiation therapy within 4 weeks prior to the first dose, except for palliative radiation (e.g., for bone metastases to control pain) that is unlikely to affect bone marrow function, which may allow inclusion 2 weeks post-radiation.
4. Patients with unstable central nervous system (CNS) metastases (those who have received treatment for brain metastases, have stable brain lesions, and have discontinued corticosteroids, anticonvulsants, or mannitol treatment for ≥2 weeks before the first dose may be considered for inclusion); patients with leptomeningeal metastases or spinal cord compression.
5. History of other primary malignancies within the past 3 years, except for malignancies that have been treated curatively with no known active disease and a low risk of recurrence, or adequately treated non-melanoma skin cancers, cervical carcinoma in situ, or papillary thyroid carcinoma.
6. Clinically significant cardiovascular diseases, including but not limited to:

   * a) Unstable angina, acute myocardial infarction, or New York Heart Association (NYHA) class II-IV heart failure;
   * b) Ventricular arrhythmias or conduction disorders requiring clinical intervention (e.g., complete left bundle branch block, third-degree atrioventricular [AV] block, or second-degree AV block);
   * c) Uncontrolled atrial fibrillation or atrial flutter;
   * d) Prolonged QTcF interval (resting mean QTcF >450 msec for men or >470 msec for women);
   * e) Left ventricular ejection fraction (LVEF) <50% on echocardiography;
   * f) Hypertension not controlled with medication.
7. • History of interstitial lung disease (ILD) or non-infectious pneumonitis.
8. • Adrenal insufficiency.
9. • Use of proton pump inhibitors, strong CYP3A4 inhibitors or inducers, or P-glycoprotein inhibitors or inducers within 7 days before the first dose.
10. • History of chronic diarrhea or diseases causing chronic diarrhea, such as Crohn's disease or irritable bowel syndrome, or any condition that might affect drug absorption (e.g., continuous diarrhea >CTCAE grade 1 within 1 week prior to the first dose).
11. • Known severe hypersensitivity to the study drug or any of its excipients.
12. • History of deep vein thrombosis, pulmonary embolism, or any other serious thromboembolic events within 6 months before the first dose, except for catheter-related or superficial venous thrombosis, or lacunar infarcts.
13. • Clinically significant gastrointestinal bleeding or hemoptysis within 3 months before the first dose, or any other significant bleeding history (e.g., pulmonary hemorrhage).
14. • Clinically significant third-space fluid accumulation (e.g., uncontrolled ascites, pleural effusion, or pericardial effusion requiring repeated drainage).
15. • Receipt of autologous transplantation within 3 months or allogeneic organ or stem cell transplantation within 6 months prior to the first dose.
16. • Active hepatitis B virus (HBV) infection (screening positive for HBsAg or anti-HBc, and HBV DNA levels above the detection limit; patients with stable disease for at least 4 weeks after antiviral therapy may be included), active hepatitis C virus (HCV) infection (positive HCV antibodies and detectable HCV RNA), human immunodeficiency virus (HIV) infection, or active syphilis infection.
17. • Active infection requiring systemic treatment within 1 week before the first dose.
18. • History of substance abuse or any condition that, in the investigator's judgment, may interfere with study participation or assessment of study results, or any unstable condition that may compromise patient safety or compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2024-12-13 (Estimated); Primary Completion 2025-12-09 (Estimated); Study Completion 2026-04-03 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 104 weeks
  The percentage of participants who achieve a complete response (CR) or partial response (PR) according to RECIST v1.1 criteria.
Maximum Tolerated Dose (MTD) | Determined at the end of the dose-escalation phase，an average of 1 year
  The highest dose at which no more than one of six participants experiences dose-limiting toxicity (DLT).
Recommended Phase II Dose (RP2D) | Determined at the end of the dose-expansion，an average of 2 years
  The dose selected for Phase II studies based on safety, tolerability, and efficacy data.

SECONDARY OUTCOMES:
Dose-Limiting Toxicities (DLTs) | At the end of Cycle 1 (each cycle is 28 days)
  The occurrence of adverse events that prevent further dose escalation.
Safety and Tolerability | From the start of treatment until 28 days after the last dose
  Assessed by the frequency, type, and severity of adverse events (AEs) and serious adverse events (SAEs) using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Peak Plasma Concentration (Cmax) | Up to approximately 30 months
  The maximum observed concentration of the drug in plasma.
Time to Reach Maximum Concentration (Tmax) | Up to approximately 30 months.
  The time at which Cmax is observed
Half-Life (t1/2) | Up to approximately 30 months
  The time required for the plasma concentration of the drug to decrease by half.

CONTACTS AND LOCATIONS:
Overall Officials: yun fan, PHD, Study Director — Zhejiang Cancer Hospital
Locations (1):
- 浙江省杭州市拱墅区半山东路1号的英文翻译为： No. 1 Banshan East Road, Gongshu District, Hangzhou, Zhejiang Province, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No